CLINICAL TRIAL: NCT03584828
Title: Comprehensive Remote Multidisciplinary Cardiac Rehabilitation Program for Patients Unable to Attend an Institution Based Program
Brief Title: Tele-Cardiac Rehabilitation Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Robert Klempfner Heart Rehabilitation Institute, Head, Cardiovascular Prevention and Rehabilitation Institute, Sheba Medical Center, Israel, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4916-18 -SMC
Record Dates: First submitted 2018-06-24; First posted 2018-07-12 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Heart Diseases
Keywords: Cardiac Rehabilitation; exercise
MeSH Terms: conditions — Heart Diseases; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-Rehabilitation - intervention (Experimental): Following the standard rehabilitation intake process the subjects in the Tele-rehaab arm will receive physiologic consultation based on clinical stress tests and clinical data passed from the physician. The Tele-rehab arm will receive an exercise prescription and execution will be assessed and periodically adjusted in accordance to data received from the wearable device. Intensity and type of exercise will be moderate and will comply with exercise recommendations provided by ESC guidelines. A dedicated application will be installed on the mobile phone for patients in the research group and they will receive a smart sports watch.
  Interventions: Behavioral: Tele Cardiac Rehabilitation
- Usual care (No Intervention): The usual care arm will receive general recommendations for a healthy and active lifestyle and community cardiologist and primary care physician according to local guidelines.

INTERVENTIONS:
Behavioral: Tele Cardiac Rehabilitation — A multidisciplinary intervention that aims to optimize structured exercise performed in the community as prescribed by rehabilitation cardiologist, cardiac care nurse, and exercise physiologist.
  Additionally, in the intervention arm, we will provide psychological support, dietary intervention and disease management services that complement the structured physical activity - all by innovative smartphone applications and smart wearable devices, thus complementing the comprehensive secondary prevention program.
  Arms: Tele-Rehabilitation - intervention

SUMMARY:
Rehabilitation programs that take place in hospitals and rehabilitation centers and all over the world are a necessary stage for returning the patients after a cardiac event to a normal functioning. However, about 70% of patients do not apply for the hospital rehabilitation programs after the heart event that they experience. The objective of this study is to evaluate and develop a multi-stage home rehabilitation program for remote rehabilitation, based on advanced technological infrastructure and complementary clinical protocols. The study population will include about 264 clinically stable patients who are eligible for cardiac rehabilitation, but for various reasons cannot get to the rehabilitation centers.

DETAILED DESCRIPTION:
Cardiac rehabilitation (CR) is an integral part of cardiovascular disease management incorporating aspects of scientifically constructed appropriate physical exercise, dietary intervention, secondary prevention by pharmacotherapy, and psychological intervention. Despite proven benefits including reduction in mortality, hospitalizations and marked improvement in well-being and function state, the current model is restrictive and requires patients' arrival to the hospital twice a week at predetermined hours. Major limitations associated with lack of participation in an in-hospital based cardiac rehabilitation program in 20-40% of eligible patients include limited transportation, time and social/family restraints, and inconvenience. Furthermore, the limited space, even in the largest rehabilitation in Israel located at Sheba Medical Center, prohibits wider availability. Leading key opinions leaders have designated cardiac-telerehabilitation as the most viable solution for the above-mentioned limitations, and several clinical studies have demonstrated safety and efficacy of this approach, including a Cochrane review and a recent meta-analysis. Nevertheless, tele-cardiac rehabilitation is not guideline recommended yet, and prospective randomized trials are necessary to better evaluate its role.

Study will enroll patients who are eligible to participate in an in-hospital cardiac rehabilitation program but are unable to participate due to one of the above-mentioned limitations, in a structured exercise and secondary prevention program in their communities. Consenting patients will undergo a baseline cardiopulmonary exercise test (CPET) followed by randomization to usual care vs. multidisciplinary intervention as described.

In addition to monitored physical activity, patients will receive nutritional and psychological counseling. This is part of a multi-professional rehabilitation program accepted by the rehabilitation center.

The study will enroll and randomize 264subjects to usual care vs. comprehensive tele-cardiac rehabilitation (TCR) with disease management services and demonstrate a greater improvement in functional capacity (O2 consumption) and improved clinical outcomes (secondary endpoints) in the TCR group.

Concomitant medications and guidelines: As indicated by national guidelines. No limitations

Study Duration: 12-month intervention period. Primary endpoint (percent change in O2 consumption) will be assessed following 3 months of intervention. Clinical event adjudication (hospitalizations, emergency department visits) will be performed throughout a 12-month period from enrollment.

Study Design: The study is an open-labeled double arm randomized prospective multi-center study designed to assess the effects of tele-CR compared to usual care in subjects that are unable to attend institution based CR despite compelling indications to CR. The intervention will be evaluated against usual care by family physician and cardiologist. The multidisciplinary program will include elements of education, nutritional and psychological interventions, monitored personalized exercise and medication titration according to the relevant national guidelines. The present sample will facilitate an evaluation of the hypothesis that tele-rehabilitation will be associated with a significant improvement in functional capacity, as assessed by the gold standard of CPET. We also hypothesize that the comprehensive intervention will also reduce clinical events, including all-cause hospitalization and death.

All subjects will undergo a detailed evaluation by rehabilitation specialist, nurse case manager, trainers and exercise physiologists. Both research arms will receive a dedicated application with a built-in pedometer and the ability to answer questionnaires.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients must meet all of the following inclusion criteria during the initial screening visit of the study (visit 1):

* A guideline-based and Israeli Health Basket approved indications for cardiac rehabilitation yet participant declines to participate in center based cardiac rehabilitation due to non-medical reasons such as: distance, service availability in subjects living are, time constraints and other logistic or sociocultural barriers
* Age ≥ 21
* Compatible smartphone (android or iOS) with internet connection
* Willing and able to comply with study protocol
* Able and willing to follow the personalized exercise prescription, use wearable technology and smartphone app, and upload data via personal smartphone

Exclusion Criteria:

Eligible patients must meet none of the following exclusion criteria:

* Any unresolved cardiac condition associated with significantly increased risk during outpatient activity (clinically significant ischemia, unresolved arrhythmia, high falling risk etc.)
* End stage \ NYHA 4 or unstable heart failure (clinical) or unresolved significant arrhythmia (i.e. Rapid atrial fibrillation)
* LVEF ≤35% without ICD \ CRTD
* Significant neurological or cognitive impairment or markedly unstable gait \ high falling risk
* Women of child-bearing potential
* ACS within 30 days prior to screening, or having undergone cardiac surgery within 30 days prior to screening
* Inability to perform a stress test due to physical limitations
* Severe angina pectoris as defined by CCS >2
* Pulmonary disease of severity greater than mild (COPD, Asthma, ILD, CTD with lung involvement) or chronic pulmonary thromboembolic disease (CTED)
* Severe orthopedic limitations
* Active myocarditis, constrictive pericarditis, restrictive or hypertrophic cardiomyopathy
* Severe Aortic or Mitral stenosis
* Significant anemia (Hb <10 mg/dl)
* Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or in the opinion of the investigator are not suitable to participate;
* Any illness which reduces life expectancy to less than 1 year from screening

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Change in METS | 6 month
  Exercise capacity change by stress test

SECONDARY OUTCOMES:
First CV hospitalization or death | 1-12 month
  Time to first cardiovascular hospitalization or death
Health status | 1-12 month
  General clinical status (worsened\ unchanged\ improved)
QOL | 1-12 month
  Assessed by validated questioner
Time alive and out of hospital | 1-12 month
Depression | 1-12 month
  Assessed by PHQ-9
Time to return to work | 1-12 month
  (if applicable)
Medication compliance | 1-12 month
  Use of guideline recommended medication and dose attained (% of target)
Fasting Glucose | 1-12 month
  levels of fasting blood glucose
Activity | 1-6 month
  average weekly steps
TCR group adherence | 1-6 month
  Percent of total exercise time at the designated target heart rate zone
TCR group sessions > 10 min adherence | 1-6 month
  Number of exercise sessions > 10 minutes per month (within target heart rate designated zone)
Lipid profile | 1-6 months
  Lipid profile dynamics
Diabetes management | 1-6 months
  HB A1C %
BMI | 1-6 months
  Change in BMI from baseline to 3 and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Cardiac Rehabilitation Institute, Tel Litwinsky, Israel